CLINICAL TRIAL: NCT06595797
Title: A Multicenter, Randomized, Double-blind, Placebo-parallel-controlled Phase II Clinical Study Evaluating the Efficacy and Safety of HRS9531 Injection in Obese Subjects With Polycystic Ovary Syndrome
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS9531-207
Record Dates: First submitted 2024-08-20; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Obese Subjects With Polycystic Ovary Syndrome (PCOS)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group 1 (Experimental)
  Interventions: Drug: HRS9531; Drug: HRS9531placebo
- Treatment group 2 (Experimental)
  Interventions: Drug: HRS9531; Drug: HRS9531placebo
- Treatment group 3 (Experimental)
  Interventions: Drug: HRS9531; Drug: HRS9531placebo

INTERVENTIONS:
Drug: HRS9531 — HRS9531
Drug: HRS9531placebo — HRS9531placebo

SUMMARY:
Randomized, double-blind, placebo-controlled study of HRS9531 in PCOS subjects

ELIGIBILITY:
Inclusion Criteria:

1. With my consent and signed informed consent, I am willing and able to complete this study in accordance with the requirements of the experimental protocol
2. Women aged 18-40 (including the threshold) on the date of signing the informed consent;
3. Patients who meet the diagnostic criteria for polycystic ovary syndrome;
4. Body mass index (BMI) ≥28 kg/m2;
5. Have controlled diet and exercise for at least 3 months, and the weight change is less than 5 kg
6. Within 2 months from the signing of the informed consent to the last drug use, there is no family planning and consent to take trial-approved contraceptive measures, and there is no egg donation plan

Exclusion Criteria:

1. Endometrial biopsy is necessary as assessed by the investigators, and the pathology of the endometrial biopsy indicates significant abnormalities
2. 12-lead electrocardiogram (ECG) results showing clinically significant abnormalities that may affect the safety of the subject, including but not limited to myocardial infarction, severe arrhythmias (e.g., supraventricular tachycardia, atrial fibrillation, atrial flutter, degree II or III atrioventricular block, etc.), and QTcF > 470 ms
3. Poor blood pressure control (with or without antihypertensive therapy) : systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg at screening
4. PHQ-9 score ≥15 points
5. The presence of endocrine disorders or medical history that may significantly affect body weight
6. Presence of other medical conditions or history that may cause hyperandrostenia or irregular menstruation
7. Presence of a history of gynecological conditions that may affect the evaluation of menstruation (including, but not limited to, history of hysterectomy, vaginal atresia, uterine adhesions)
8. Abnormal uterine bleeding for reasons other than PCOS or unexplained abnormal uterine bleeding occurred within 6 months
9. Endometrium-related surgery within 1 year indicated significant pathological abnormalities of endometrial tissue, and safety risks were assessed by researchers
10. History of pregnancy, miscarriage, childbirth or breastfeeding within 6 months
11. Have any disease or history that affects gastric empty. such as gastric bypass surgery, pyloric stenosis, etc., long-term use of drugs that directly affect gastrointestinal motility, serious gastrointestinal disease (such as active peptic ulcer, inflammatory bowel disease, etc.), or have undergone gastrointestinal surgery (except surgery that has no significant effect on gastrointestinal motility), Such as gastrointestinal polypectomy, appendectomy and hemorrhoid surgery);
12. A history or disease of acute or chronic pancreatitis or pancreatic injury; Patients with a history of acute cholecystitis or symptomatic/treatable gallbladder disease (except those who had previously undergone cholecystectomy and were deemed eligible by the investigator to be enrolled);
13. History or family history of medullary thyroid carcinoma (MTC) or multiple endocrine adenomatosis type 2 (MEN2);
14. Severe infection, severe trauma, or major or major surgery in the previous 6 months
15. A history of severe cardiovascular and cerebrovascular disease, including decompensated heart failure (New York Heart Association ratings III and IV), unstable angina pectoris, stroke or transient ischemic attack, myocardial infarction, severe arrhythmia, or coronary bypass grafting or percutaneous coronary intervention within the previous 6 months;
16. Any organ-system malignancy within the previous 5 years, regardless of evidence of local recurrence or metastasis, except cured local basal cell carcinoma of the skin, cervical carcinoma in situ, and prostate carcinoma in situ;
17. Present or suspected depression, anxiety disorder, bipolar disorder, suicidal tendencies, schizophrenia, or other more serious mental illness
18. A known or suspected history of alcohol and/or drug abuse or drug use
19. A history of acute or chronic hepatitis, or other serious liver disease other than alcoholic fatty liver disease;
20. A history of unstable or rapidly progressing kidney disease or end-stage kidney disease
21. Autoimmune disease is present and systemic glucocorticoid therapy or immunosuppressive therapy is planned for the study period;
22. Participated in a clinical trial of any drug or medical device within the previous 3 months, defined as signing informed consent and using the investigational drug (including placebo) or the investigational medical device; Or is still in the trial drug within 5 half-lives (whichever is older);
23. Those who have donated blood or lost blood ≥400 mL in the previous 3 months, or received blood transfusion
24. Surgery is planned during the trial period (except for minor surgery that the investigator believes will not affect the trial);
25. Mentally incapacitated or speech-impaired subjects are unable to fully understand or participate in the test process;
26. Researchers and relevant staff of the research Centre or others directly involved in the implementation of the programme, as well as members of their immediate family (e.g. spouse, legal partner, parents, children or siblings); Hengrui company staff;
27. There are circumstances (medical, psychological, social or geographical factors, etc.) that, in the investigator's judgment, affect the subject's safety or any other conditions that interfere with the evaluation of the test results.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percentage change in body weight from baseline at 32 weeks of treatment | 0week, 4week ,8week, 12week, 16week, 20week , 24week, 28week, 32week

SECONDARY OUTCOMES:
Proportion of subjects with regular menstruation at 32 weeks of treatment | 0week, 4week ,8week, 12week, 16week, 20week , 24week, 28week, 32week
Change in spontaneous menstrual frequency ratio from baseline at 32 weeks of treatment | 0week, 4week ,8week, 12week, 16week, 20week , 24week, 28week, 32week
Proportion of subjects who ovulated regularly after 32 weeks of treatment | 0week, 4week ,8week, 12week, 16week, 20week , 24week, 28week, 32week
Proportion of subjects with weight loss of ≥5%, ≥10%, ≥15%, ≥20% from baseline at 32 weeks of treatment | 0week, 4week ,8week, 12week, 16week, 20week , 24week, 28week, 32week
BMI changes relative to baseline after 32 weeks of administration; | 0week, 4week ,8week, 12week, 16week, 20week , 24week, 28week, 32week
Changes in waist circumference (WC) from baseline after 32 weeks of administration | 0week, 4week ,8week, 12week, 16week, 20week , 24week, 28week, 32week
Proportion of subjects with at least 3 menstrual cycles of 21-35 days after 12-32 weeks of treatment; | 0week, 4week ,8week, 12week, 16week, 20week , 24week, 28week, 32week
Changes in total testosterone (TT)from baseline after 32 weeks of administration | 0week, 12week, 24week, 32week
Changes in sex hormone binding globulin (SHBG)from baseline after 32 weeks of administration | 0week, 12week, 24week, 32week
Changes in free testosterone index (FAI),from baseline after 32 weeks of administration | 0week, 12week, 24week, 32week
Changes in anti-Miller tube hormone (AMH),from baseline after 32 weeks of administration | 0week, 12week, 24week, 32week
Changes in follicle stimulating hormone (FSH),from baseline after 32 weeks of administration | 0week, 12week, 24week, 32week
Changes in luteinizing hormone (LH)from baseline after 32 weeks of administration | 0week, 12week, 24week, 32week
Changes in LH/FSH;from baseline after 32 weeks of administration | 0week, 12week, 24week, 32week
Changes in fasting plasma glucose (FPG)from baseline after 32 weeks of administration | 0week, 12week, 24week, 32week
Changes in fasting serum insulin (FINS),from baseline after 32 weeks of administration | 0week, 12week, 24week, 32week
Changes in insulin resistance index (HOMA-IR)from baseline after 32 weeks of administration | 0week, 12week, 24week, 32week
Changes in triglycerides from baseline after 32 weeks of administration | 0week, 12week, 24week, 32week
Changes in total cholesterol (TC),from baseline after 32 weeks of administration | 0week, 12week, 24week, 32week
Changes in, low density lipoprotein cholesterol (LDL-C)from baseline after 32 weeks of administration | 0week, 12week, 24week, 32week
Changes in high density lipoprotein cholesterol (HDL-C)from baseline after 32 weeks of administration | 0week, 12week, 24week, 32week
Changes in blood pressure from baseline | 0week, 4week,12week, 24week, 32week
Adverse events, | 0week, 4week ,8week, 12week, 16week, 20week , 24week, 28week, 32week

IPD SHARING:
Plan to Share IPD: Undecided